CLINICAL TRIAL: NCT04818983
Title: The Exploratory Study to Evaluate Biomarkers in Prospective Multicenter Observational Study of Atezolizumab Combination Therapy in Patients With Unresectable, Advanced and Recurrent Non-small Cell Lung Cancer or Extensive Disease Small Cell Lung Cancer (J-TAIL-2)
Brief Title: The Biomarker Exploratory Study in Prospective Multicenter Observational Study of Atezolizumab Combination Therapy in Lung Cancer (J-TAIL-2)
Status: Completed | Type: Observational
Sponsor: Chugai Pharmaceutical (Industry)
Collaborators: Japan Lung Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: J-TAIL-2 biomarkers
Record Dates: First submitted 2021-03-19; First posted 2021-03-26 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Non-small Cell Lung Cancer; Extensive Disease Small Cell Lung Cancer
Keywords: Atezolizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The biomarkers which enable to select the appropriate patient in atezolizumab combination therapy are exploratory examined with the 3 methods below.
  * Analysis of PD-L1 SNPs
  * Comprehensive analysis of plasma protein expression
  * Analysis of the immune microenvironment of small cell lung cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NSCLC cohort: Patients with locally advanced or metastatic non-small cell lung cancer who are planning to provide atezolizumab combination therapy as the most appropriate medical care
- ED-SCLC cohort: Patients with extensive disease small cell lung cancer who are planning to provide atezolizumab combination therapy as the most appropriate medical care

SUMMARY:
This study is implemented in association with the study "J-TAIL-2" ; prospective multicenter observational study of atezolizumab in patients with unresectable, locally advanced or metastatic non-small cell lung cancer, UMIN study ID: UMIN000041263, to evaluate biomarkers for selection of appropriate patients in treatment with atezolizumab combination therapy.

ELIGIBILITY:
Inclusion Criteria:

Inclusion/exclusion criteria of J-TAIL-2 study is to be applied.

<non-small cell lung cancer cohort>

1. Patients 20 years of age or older at the time of signed consent.
2. Patients with unresectable, advanced and recurrent non-small cell lung cancer.
3. Patients who are scheduled to start atezolizumab combination therapy in clinical practice, based on the atezolizumab package insert and the Optimal Clinical Use Guideline.
4. Patients who signed informed consent form before enrolling the study. The consent from a legally acceptable representative is required for the patients with uncertain capacity of judgments.

<extensive disease small cell lung cancer cohort>

1. Patients 20 years of age or older at the time of signed consent.
2. Patients with extensive disease small cell lung cancer.
3. Patients who are scheduled to start atezolizumab combination therapy in clinical practice, based on the atezolizumab package insert and the Optimal Clinical Use Guideline.
4. Patients who signed informed consent form before enrolling the study. The consent from a legally acceptable representative is required for the patients with uncertain capacity of judgments. However, the samples of dead cases can be used for the analysis of immune microenvironment of small cell lung cancer by disclosing information on this study.

Exclusion Criteria:

<non-small cell lung cancer cohort>

1. Patients who are unsuitable for enrolment into the study by the investigator's judgment.

<extensive disease small cell lung cancer cohort>

1. Patients who are unsuitable for enrolment into the study by the investigator's judgment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are planning to provide atezolizumab combination therapy as the most appropriate medical care for patients and who meet the Eligibility criteria at registration.
Sampling Method: Non-Probability Sample
Enrollment: 470 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Correlation between PD-L1 SNP and atezolizumab combination therapy | Baseline
Correlation between rate of change in plasma protein expression level and atezolizumab combination therapy | Baseline, Predose of cycle 2 (each cycle is 21 days), and when immune-related adverse event occurs (through study completion, an average of 2 years 5 months)
Correlation between an immune microenvironment of small cell lung cancer and atezolizumab combination therapy | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Akihiko GENMA, Principal Investigator — Nippon Medical School
Locations (95):
- Japan (95):
  - Hyogo Cancer Center, Akashi
  - Asahikawa Medical University Hospital, Asahikawa
  - National Hospital Organization Asahikawa Medical Center, Asahikawa
  - Juntendo University Hospital, Bunkyō City
  - Nippon Medical School Hospital, Bunkyō City
  - Tokyo Medical And Dental University, Medical Hospital, Bunkyō City
  - Chiba University Hospital, Chiba
  - National Cancer Center Hospital, Chūōku
  - Fukuoka University Hospital, Fukuoka
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - National Hospital Organization Okinawa National Hospital, Ginowan
  - National Hospital Organization Himeji Medical Center, Himeji
  - Kansai Medical University Hospital, Hirakata
  - Hirosaki University Hospital, Hirosaki
  - Hiroshima University Hospital, Hiroshima
  - Aso Iizuka Hospital, Iizuka
  - Nippon Medical School Chiba Hokusoh Hospital, Inzai
  - Tokai University Hospital, Isehara
  - Teikyo University Hospital, Itabashi-Ku
  - Itami City Hospital, Itami
  - National Hospital Organization Iwakuni Clinical Center, Iwakuni
  - Shimane University Hospital, Izumo
  - Kagawa University Hospital, Kagawa
  - Kagoshima University Hospital, Kagoshima
  - Kanazawa University Hospital, Kanazawa
  - Kasukabe Medical Center, Kasukabe
  - Hospital of the University of Occupational and Envioronmental Health, Kitakyushu
  - Kitakyushu Municipal Medical Center, Kitakyushu
  - Japan Anti-Tuberculosis Association Fukujuji Hospital, Kiyose
  - Kobe Minimally Invasive Cancer Center, Kobe
  - Kobe University Hospital, Kobe
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Kōtoku
  - Kurume University Hospital, Kurume
  - Kyoto City Hospital, Kyoto
  - Kyoto University Hospital, Kyoto
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Shinshu University Hospital, Matsumoto
  - Matsusaka Municipal Hospital, Matsusaka
  - National Hospital Organization Tokyo Medical Center, Meguro-Ku
  - The Jikei University Hospital, Minatoku
  - Miyazaki Prefectural Miyazaki Hospital, Miyazaki
  - Aichi Medical University Hospital, Nagakute
  - Nagasaki University Hospital, Nagasaki
  - Aichi Cancer Center, Nagoya
  - Nagoya City University Hospital, Nagoya
  - Nagoya University Hospital, Nagoya
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - Miyagi Cancer Center, Natori
  - Niigata Cancer Center Hospital, Niigata
  - Niigata University Medical and Dental Hospital, Niigata
  - The Hospital of Hyogo College of Medicine, Nishinomiya
  - Obihiro Kosei Hospital, Obihiro
  - Japanese Red Cross Okayama Hospital, Okayama
  - Kawasaki Medical School General Medical Center, Okayama
  - Okayama Rosai Hospital, Okayama
  - Okayama University Hospital, Okayama
  - Osaka City General Hospital, Osaka
  - Osaka General Medical Center, Osaka
  - Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Ōsaka-sayama
  - Gunma Prefectural Cancer Center, Ōta-ku
  - Shiga University of Medical Science Hospital, Ōtsu
  - Saitama medical university International medical Center, Saitama
  - Saitama Prefectural Cancer Center, Saitama
  - Saitama Red Cross Hospital, Saitama
  - National Hospital Organization Kinki-Chuo Chest Medical Center, Sakai
  - Hokkaido University Hospital, Sapporo
  - Teine Keijinkai Hospital, Sapporo
  - Sendai Kousei Hospital, Sendai
  - Tohoku Medical And Pharmaceutical University Hospital, Sendai
  - Tohoku University Hospital, Sendai
  - Showa University Hospital, Shinagawa-Ku
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-Ku
  - Keio University Hospital, Shinjuku-Ku
  - Iwate Medical University Hospital, Shiwa-gun
  - Osaka University Hospital, Suita
  - Saiseikai Suita Hospital, Suita
  - Kagawa Prefectural Central Hospital, Takamatsu
  - JA Toyama Kouseiren Takaoka Hospital, Takaoka
  - Takarazuka City Hospital, Takarazuka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki
  - Tenri Hospital, Tenri
  - Dokkyo Medical University Hospital, Tochigi
  - Tokushima Prefectural Central Hospital, Tokushima
  - Tokushima University Hospital, Tokushima
  - Toyama Prefectural Central Hospital, Toyama
  - Fujita Health University Hospital, Toyoake
  - National Hospital Organization Yamaguchi-Ube Medical Center, Ube
  - Wakayama Medical University Hospital, Wakayama
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama
  - Yokohama City University Hospital, Yokohama
  - Tottori University Hospital, Yonago
  - Oita University Hospital, Yufu

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the end of the study